CLINICAL TRIAL: NCT01380327
Title: A Biomarker-Based Pilot Study of Cockroach Sublingual Immunotherapy in Cockroach Sensitive Children With Asthma and/or Perennial Allergic Rhinitis
Brief Title: Biomarkers of Cockroach Sublingual Immunotherapy 2
Acronym: BioCSI-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ICAC-17
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2014-05-30 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Asthma; Perennial Allergic Rhinitis
Keywords: cockroach; immunotherapy; sublingual immunotherapy (SLIT); inner city asthma
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cockroach Sublingual Immunotherapy (SLIT) - Low Dose (Experimental): Glycerinated German cockroach (Blatella germanica) allergen extract administered sublingually with a maximally tolerated dose of 420 microliters daily
  Interventions: Biological: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose
- Placebo (Placebo Comparator): Placebo administered sublingually not to exceed the maximally tolerated dose of either 1.) 420 microliters daily (placebo - low dose randomization) or 2.) 840 microliters twice daily (placebo - high dose randomization)
  Interventions: Other: Placebo
- Cockroach Sublingual Immunotherapy (SLIT) - High Dose (Experimental): Glycerinated German cockroach (Blatella germanica) allergen extract administered sublingually with a maximally tolerated dose of 840 microliters taken twice daily
  Interventions: Biological: Cockroach Sublingual Immunotherapy (SLIT) - High Dose

INTERVENTIONS:
Biological: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose — Participants are randomized to receive daily doses of glycerinated German cockroach (Blattella germanica) allergenic extract formulated in 50% glycerin at a concentration of 1:20 weight per volume [w/v] placed under the tongue (sublingual route) to dissolve. The treatment course and study duration was 3 months. Note: The extract was also administered during the preliminary dosing visits, up to three escalating doses, or until the maximum study dose (420 microliters, 1:20 w/v) was achieved.
  Other Names: Blattella germanica
  Arms: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose
Other: Placebo — Participants are randomized to receive either daily (low dose) or twice-daily (high dose) placebo treatment placed under the tongue (sublingual route) to dissolve. The treatment course and study duration was 3 months. Note: The placebo was also administered during the preliminary dosing visits, up to three or seven escalating doses, or until the maximum study dose (420 or 840 microliters, 1:20 weight per volume [w/v]) was achieved.
  Other Names: German cockroach (Blattella germanica) placebo
  Arms: Placebo
Biological: Cockroach Sublingual Immunotherapy (SLIT) - High Dose — Participants are randomized to receive twice-daily doses of glycerinated German cockroach (Blattella germanica) allergenic extract formulated in 50% glycerin at a concentration of 1:20 weight per volume [w/v] placed under the tongue (sublingual route) to dissolve. The treatment course and study duration was 3 months. Note: The extract was also administered during the preliminary dosing visits, up to seven escalating doses, or until the maximum study dose (840 microliters, 1:20 w/v) was achieved.
  Other Names: Blattella germanica
  Arms: Cockroach Sublingual Immunotherapy (SLIT) - High Dose

SUMMARY:
This trial is a follow-up study of the ICAC-12 Phase I/II trial (NCT00829985), and is designed to study biomarkers of the immune response to allergen immunotherapy and the safety of this therapy in a pediatric population.

DETAILED DESCRIPTION:
Over the past two decades, scientific evidence has shown that the combination of cockroach allergy and cockroach exposure is one of the most important factors contributing to the dramatic increase in asthma morbidity seen in inner city children with asthma. Therefore, a major goal of the National Institute of Allergy and Infectious Diseases (NIAID) Inner City Asthma Consortium (ICAC) is ultimately to conduct a large multi-center trial of cockroach sublingual immunotherapy (SLIT) in inner-city asthma. As a step toward achieving this goal, ICAC is conducting a clinical trial comparing two doses of glycerinated German cockroach (Blattella germanica) allergenic extract to placebo, administered under the tongue (sublingual).

ELIGIBILITY:
Inclusion Criteria:

* Have a history of perennial allergic rhinitis, asthma, or both, before study entry. For those with asthma:

  1. a diagnosis of asthma will be defined as a report by the participant that they have had a clinical diagnosis of asthma made by a physician over a year ago
  2. the participant's asthma must be well controlled as defined by: ii. a forced expiratory volume at one second (FEV1) greater than or equal to 80% predicted value with or without controller medication ii. albuterol use for no more than 3 days per week in each of the previous 2 weeks for asthma symptoms (not including exercise prophylaxis)
* Are sensitive to German cockroach (Blattella germanica) as documented by a positive (>/=3 mm greater than negative control) skin prick test result and detectable German cockroach specific IgE (>/=0.35 kUA/L)
* Have no known contraindications to therapy with glycerinated German cockroach allergenic extract or placebo
* Parent or legally authorized representative (LAR) of child is willing to sign the written Informed Consent prior to initiation of any study procedure

Exclusion Criteria:

* Are pregnant or lactating. Females must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral, subcutaneous, mechanical, or surgical contraception)
* Cannot perform spirometry or peak flow at screening
* Have an asthma severity classification at recruitment of severe persistent, using the National Asthma Education and Prevention Program (NAEPP) classification, as evidenced by at least one of the following:

  1. requires a dose of greater than 500 mcg of fluticasone per day or the equivalent of another inhaled corticosteroid
  2. have received more than 2 courses of oral or parenteral corticosteroids within the last 12 months
  3. have been treated with depot steroids within the last 12 months
  4. have been hospitalized for asthma within the 6 months prior to recruitment
  5. have had a life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within 2 years prior to recruitment
* Do not have access to a phone (needed for scheduling appointments)
* Have received allergen immunotherapy in the last 12 months prior to recruitment or who plan to initiate or resume allergen immunotherapy during the study
* Have previously been treated with anti-IgE therapy within 1 year of recruitment
* Have received an investigational drug in the 30 days prior to recruitment or who plan to use an investigational drug during the study
* Have in the last 3 months prior to recruitment experienced on average >/=1 day per week any of the symptoms below:

  1. nausea or vomiting
  2. abdominal pain or cramps severe enough to interfere with daily activities (excluding those associated with menstruation).
  3. diarrhea
* Refuse to sign the Epinephrine Auto-injector Training Form

Participants who meet any of the following criteria are not eligible for enrollment and may not be reassessed. Participants are ineligible if they:

* Do not primarily speak English
* Plan to move from the area during the study period
* Have a history of idiopathic anaphylaxis or anaphylaxis grade 2 or higher
* Have unstable angina, significant arrhythmia, uncontrolled hypertension, history of autoimmune disease, or other chronic or immunological diseases that in the opinion of the investigator might interfere with the evaluation of the investigational agent or pose additional risk to the patient (e.g., gastrointestinal disease, gastroesophageal reflux disease, chronic infections, scleroderma, hepatic, and gallbladder disease)
* Are using tricyclic antidepressants or beta-adrenergic blocker drugs (either oral and/or topical route[s] of administration)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Study Chair — Johns Hopkins University
Locations (5):
- United States (5):
  - Children's Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Wood RA, Togias A, Wildfire J, Visness CM, Matsui EC, Gruchalla R, Hershey G, Liu AH, O'Connor GT, Pongracic JA, Zoratti E, Little F, Granada M, Kennedy S, Durham SR, Shamji MH, Busse WW. Development of cockroach immunotherapy by the Inner-City Asthma Consortium. J Allergy Clin Immunol. 2014 Mar;133(3):846-52.e6. doi: 10.1016/j.jaci.2013.08.047. Epub 2013 Nov 1. PMID 24184147
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five NIAID ICAC sites in the United States recruited the targeted number of study participants who fulfilled entry criteria between May 2011 and February 2012. Of the ninety-nine subjects enrolled in the study, eighty-nine achieved the milestone of randomization and are included in the Participant Flow: Overall Study Results Section.
Groups:
- Cockroach Sublingual Immunotherapy (SLIT) - High Dose: Participants received twice-daily doses of glycerinated German cockroach (Blattella germanica) allergenic extract formulated in 50% glycerin at a concentration of 1:20 weight per volume [w/v] placed under the tongue (sublingual route) to dissolve. The treatment course and study duration was 3 months. Note: The extract was also administered during the preliminary dosing visits, up to seven escalating doses, or until the maximum study dose (840 microliters, 1:20 w/v) was achieved.
- Cockroach Sublingual Immunotherapy (SLIT) - Low Dose: Participants received daily doses of glycerinated German cockroach (Blattella germanica) allergenic extract formulated in 50% glycerin at a concentration of 1:20 weight per volume [w/v] placed under the tongue (sublingual route) to dissolve. The treatment course and study duration was 3 months. Note: The extract was also administered during the preliminary dosing visits, up to three escalating doses, or until the maximum study dose (420 microliters, 1:20 w/v) was achieved.
- Placebo: Participants received daily (placebo-low dose) or twice-daily (placebo - high dose) doses of placebo placed under the tongue (sublingual route) to dissolve. The treatment course and study duration was 3 months. Note: The placebo was also administered during the preliminary dosing visits, up to three or seven escalating doses, or until the maximum study dose (420 or 840 microliters, 1:20 weight per volume [w/v]) was achieved.
Period: Overall Study
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Started | 30 (Number in intent-to-treat having reached maximum tolerated dose with =/> 1 one post-baseline measure) | 31 (Number in intent-to-treat having reached maximum tolerated dose with =/> 1 one post-baseline measure) | 28 (Number in intent-to-treat having reached maximum tolerated dose with =/> 1 one post-baseline measure)
Completed | 27 | 28 | 21
Not Completed | 3 | 3 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Protocol Violation | 3 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Housing situation precluded ability to k | 0 | 0 | 1
Not completed — Questionable onset of epilepsy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 28 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (3.6) | 11.0 (3.3) | 10.8 (3.7) | 10.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 26
  Male | 21 | 22 | 20 | 63
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 28 | 89
German Cockroach-Specific Serum Immunoglobulin E (IgE) Levels [Median (Full Range); unit: kU/L] | 6.7 [0.4 to 349.0] | 4.9 [0.4 to 174.0] | 9.2 [0.4 to 98.6] | 6.4 [0.4 to 349.0]
German Cockroach-Specific Serum Immunoglobulin G (IgG) Levels [Median (Full Range); unit: mg/mL] | 4.1 [2.0 to 33.8] | 4.3 [2.0 to 20.6] | 5.1 [2.0 to 24.9] | 4.5 [2.0 to 33.8]
German Cockroach-Specific Serum Immunoglobulin Subclass 4 (IgG4) Levels [Median (Full Range); unit: mg/mL] | 0.1 [0.0 to 7.5] | 0.1 [0.0 to 3.5] | 0.5 [0.0 to 2.6] | 0.2 [0.0 to 7.5]
German Cockroach-Specific IgE Fragment Antibody Binding (FAB) Activity [Median (Full Range); unit: Percent antibody binding] | 84.9 [5.0 to 426.4] | 78.3 [6.2 to 421.7] | 80.8 [16.9 to 201.5] | 81.5 [5.0 to 426.4]
German Cockroach Prick Skin Test Wheal Size [Median (Full Range); unit: mm] | 5.0 [3.0 to 12.0] | 5.0 [3.5 to 12.0] | 5.8 [4.0 to 11.5] | 5.3 [3.0 to 12.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in German Cockroach-Specific Serum IgE Over Time
Description: Outcome is the ratio of geometric means for baseline versus post-baseline German cockroach-specific serum IgE. This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 3 months of treatment
Population: Intent-to-treat population with complete data.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Number analyzed (Participants) | 30 | 30 | 28
Ratio | 2.0 [1.6 to 2.5] | 2.7 [2.2 to 3.3] | 1.2 [1.0 to 1.5]
Statistical Analysis 1: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - High Dose vs Placebo; Analysis compared cockroach SLIT -high dose, Placebo - high dose; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Risk Ratio (RR) = 1.7, 95% CI 2-sided [1.2 to 2.3] — Estimated value & associated CI is the ratio of change (baseline to post-baseline) in placebo group (denominator=1.18) vs. high dose group (numerator=1.98)
Statistical Analysis 2: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose vs Placebo; Analysis compared cockroach SLIT - low dose, placebo - low dose; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Risk Ratio (RR) = 2.3, 95% CI 2-sided [1.7 to 3.1] — Estimated value & associated CI is the ratio of change (baseline to post-baseline) in placebo group (denominator=1.18) vs. low dose group (numerator=2.69)

2. Secondary Outcome: Change in German Cockroach-Specific Serum IgG Over Time
Description: Outcome is the ratio of geometric means for baseline versus post-baseline German cockroach-specific serum immunoglobulin G (IgG). This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 3 months of treatment
Population: Intent-to-treat population with complete data.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Number analyzed (Participants) | 30 | 31 | 28
Ratio | 1.3 [1.2 to 1.4] | 1.1 [1.1 to 1.2] | 1.0 [1.0 to 1.1]
Statistical Analysis 1: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - High Dose vs Placebo; Analysis compared cockroach SLIT - high dose, placebo - high dose; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Risk Ratio (RR) = 1.3, 95% CI 2-sided [1.1 to 1.4] — Estimated value & associated CI is the ratio of change (baseline to post-baseline) in placebo group (denominator=1.04) vs. high dose group (numerator=1.32)
Statistical Analysis 2: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose vs Placebo; Analysis compared cockroach SLIT - low dose, placebo - low dose; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis; Risk Ratio (RR) = 1.1, 95% CI 2-sided [1.0 to 1.2] — Estimated value & associated CI is the ratio of change (baseline to post-baseline) in placebo group (denominator=1.04) vs. low dose group (numerator=1.14)

3. Secondary Outcome: Change in German Cockroach-Specific Serum IgG4 Over Time
Description: Outcome is the ratio of geometric means for baseline versus post-baseline German cockroach-specific serum immunoglobulin subclass 4 (IgG4). This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 3 months of treatment
Population: Intent-to-treat population with complete data.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Number analyzed (Participants) | 29 | 30 | 27
Ratio | 1.6 [1.2 to 2.1] | 1.5 [1.1 to 1.9] | 1.0 [0.8 to 1.4]
Statistical Analysis 1: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - High Dose vs Placebo; Analysis compared cockroach SLIT - high dose, placebo - high dose; Test type: Superiority or Other; p = 0.06, Mixed Models Analysis; Risk Ratio (RR) = 1.5, 95% CI 2-sided [1.0 to 2.4] — Estimated value and associated CI is the ratio of change (baseline to post-baseline) in placebo group (denominator=1.03) vs. high dose group (numerator=1.57)
Statistical Analysis 2: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose vs Placebo; Analysis compared cockroach SLIT - low dose, placebo - low dose; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis; Risk Ratio (RR) = 1.4, 95% CI 2-sided [0.9 to 2.2] — Estimated value & associated CI is the ratio of change (baseline to post-baseline) in placebo group (denominator=1.03) vs. low dose group (numerator=1.45)

4. Secondary Outcome: Change in IgE Fragment Antibody Binding (FAB) Activity Over Time
Description: Outcome is change in mean IgE FAB activity level from baseline to post-baseline (status post 3 months of treatment). Serum from cockroach sublingual immunotherapy (SLIT)-treated participants were analyzed to determine if treatment inhibits in-vitro cockroach SLIT, using the per protocol allergenic extract doses. This result is an indicator of immune modulation over time, however its clinical significance is unclear.(Reference: Shamji MH et al. The IgE-facilitated allergen binding (FAB) assay: validation of a novel flow-cytometric based method for the detection of inhibitory antibody responses. J Immunol Methods 2006;317(1-2): 71-9).
Time Frame: Baseline through 3 months of treatment
Population: Intent-to-treat population with complete data.
Measure: Mean (95% Confidence Interval); unit: Percent antibody binding
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Number analyzed (Participants) | 30 | 28 | 24
Percent antibody binding | -7.2 [-20.8 to 6.5] | 19.2 [5.3 to 33.2] | 5.7 [-9.5 to 20.9]
Statistical Analysis 1: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - High Dose vs Placebo; Analysis compared cockroach SLIT - high dose, placebo - high dose; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis; Treatment effect = -12.9, 95% CI 2-sided [-33.2 to 7.5] — Estimated value& associated CI is the treatment effect: baseline to post-baseline change in measurement in high dose group (-7.2) minus baseline to post-baseline change in measurement in placebo group (5.7)
Statistical Analysis 2: Comparison: Cockroach Sublingual Immunotherapy (SLIT) - Low Dose vs Placebo; Analysis compared cockroach SLIT - low dose, placebo - low dose; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis; Treatment effect = 13.5, 95% CI 2-sided [-7.1 to 34.1] — Estimated value& associated CI is the treatment effect: baseline to post-baseline change in measurement in high dose group (19.2) minus baseline to post-baseline change in measurement in placebo group (5.7)

5. Secondary Outcome: Percent of Participants With the Occurrence of Adverse Events (AEs)
Description: Percent of participants who experienced at least one AE.
Time Frame: Participant enrollment to end of study (up to 3 months post-baseline)
Measure: Number; unit: Percentage of population
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Number analyzed (Participants) | 34 | 33 | 32
Percentage of population | 59 | 76 | 66

ADVERSE EVENTS:
Time Frame: Participant enrollment to end of study (up to 3 months post-baseline)
Description: This study graded the severity of adverse events experienced by the study participant according to criteria set forth in the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 3.0 (June 10, 2003)
Groups:
- Cockroach Sublingual Immunotherapy (SLIT) - High Dose: Participants with German cockroach allergy and mild to moderate asthma, rhinitis, or both self-administered concentrated (1:20 weight per volume [w/v]) twice-daily doses of glycerinated German cockroach allergenic extract (50% glycerin) placed under the tongue (sublingually) to dissolve. The treatment course and study duration was 3 months. Note: The extract was also administered during the preliminary dosing visits, up to seven escalating doses, or until the maximum study dose (840 microliters, 1:20 w/v) was achieved.
- Cockroach Sublingual Immunotherapy (SLIT) - Low Dose: Participants with German cockroach allergy and mild to moderate asthma, rhinitis, or both self-administered concentrated (1:20 weight per volume [w/v]) daily doses of glycerinated German cockroach allergenic extract (50% glycerin) placed under the tongue (sublingually) to dissolve. The treatment course and study duration was 3 months. Note: The extract was also administered during the preliminary dosing visits, up to three escalating doses, or until the maximum study dose (420 microliters, 1:20 w/v) was achieved.
- Placebo: Participants with German cockroach allergy and mild to moderate asthma, rhinitis, or both self-administered daily or twice-daily doses of placebo placed under the tongue (sublingually) to dissolve. The treatment course and study duration was 3 months. Note: The placebo was also administered during the preliminary dosing visits, up to three or seven escalating doses, or until the maximum study dose (420 or 840 microliters, 1:20 weight per volume [w/v]) was achieved.
Arm/Group | Cockroach Sublingual Immunotherapy (SLIT) - High Dose | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 2/32
Other Adverse Events (participants affected / at risk) | 20/34 | 25/33 | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cockroach Sublingual Immunotherapy (SLIT) - High Dose (N=34) | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose (N=33) | Placebo (N=32)
Renal disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cockroach Sublingual Immunotherapy (SLIT) - High Dose (N=34) | Cockroach Sublingual Immunotherapy (SLIT) - Low Dose (N=33) | Placebo (N=32)
Ear pruritus (Ear and labyrinth disorders) | 3 (3) | 4 (8) | 1 (1)
Eye pruritus (Eye disorders) | 3 (3) | 4 (4) | 5 (10)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (3) | 2 (3)
Oral pruritus (Gastrointestinal disorders) | 2 (3) | 4 (5) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Tongue pruritus (Gastrointestinal disorders) | 1 (1) | 5 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (9) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 4 (4) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 10 (14) | 6 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (7) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (8) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No